CLINICAL TRIAL: NCT02650375
Title: A Phase Ib Clinical Study of the Tolerance, Safety and Preliminary Efficacy Observation of Single-/Multiple- Doses of Metatinib Tromethamine Tablets in Patients With Advanced or Metastatic Solid Tumor
Brief Title: Study of Metatinib Tromethamine Tablet
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-128-I-02
Record Dates: First submitted 2015-11-10; First posted 2016-01-08 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Advanced or Metastatic Gastric Cancer; Advanced or Metastatic Liver Cancer; Advanced or Metastatic CRC; Advanced or Metastatic Non Squamous NSCLC
MeSH Terms: conditions — Stomach Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metatinib Tromethamine (Experimental)
  Interventions: Drug: Metatinib Tromethamine

INTERVENTIONS:
Drug: Metatinib Tromethamine — Patients receive Metatinib orally 200mg once daily (QD) or 100mg twice daily (BID) until disease progression or unacceptable toxicity occurred.

SUMMARY:
This is an open-label, multicenter study designed to assess the safety, tolerability, preliminary efficacy and pharmacokinetics of Metatinib Tromethamine tablet in patients with advanced or metastatic gastric cancer, liver cancer, colorectal cancer,or con squamous NSCLC. Patients receive Metatinib orally 200mg once daily (QD) or 100mg twice daily (BID) until disease progression or unacceptable toxicity occurred. The study will determine whether MET gene mutation, amplification, as well as MET protein overexpression in tumor tissue correlate with treatment efficacy and clinical outcome. The potential PD biomarker for Metatinib will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic gastric cancer or colorectal cancer who progress after second-line therapy or the above treatment protocol, or patients with advanced or metastatic hepatocellular carcinoma who progress after first-line chemotherapy, interventional therapy or targeted therapy shall be verified by histology or cytology; or patients with advanced or metastatic non-squamous non-small cell lung cancer who cannot be operated or fail to first-line therapy shall be verified by histology or cytology;
* MET gene amplification or protein overexpression(IHC ≥2+）,or exon-14 skipping;
* At least one measurable lesion (RECIST 1.1 );
* At least 4 weeks from the last chemotherapy, radiotherapy or anti-tumor biological products treatment; at least 8 weeks from the last anti-tumor antibody products treatment; at least 6 weeks from the last dose of nitrosourea, mitomycin C or doxorubicin;
* At least 4 weeks from major surgery or trauma, and the wound should fully heal; at least 1 week from minor surgery or trauma (i.e. tissue biopsy or fine needle aspiration);
* Toxicity from previous treatment has to restore to ≤ grade 1, baseline or irreversible (NCI CTC4.0);
* ECOG performance status 0-1;
* Life expectancy ≥3 months;
* Adequate hematologic function: ANC≥1.5×10^9 /L, HB≥90g/L(blood transfusion allowed), PLT≥100×10^9/L;
* Adequate hepatic function: ALT≤3×ULN, AST≤3×ULN, TBIL≤2×ULN(patients with liver metastases or liver cancer ALT≤5×ULN, AST≤5×ULN, TBIL≤2×ULN), Child-Pugh score≤7;
* Adequate renal function: uric acid<500μmol/L, creatinine<1.7mg/dL, proteinuria≤2＋or≤2g/24h , GFR≥60 ml/min/1.73m^2;
* PT-INR/APTT≤1.5×ULN, Serum sodium, potassium, calcium, magnesium levels ≤1×ULN(NCI-CTC 4.0);
* Patients signed written informed consent;
* Willingness and capability to comply with protocol requirement and well communicate with investigators.

Exclusion Criteria:

* Severe, uncontrolled medical disorders or active infection, including but not limited to HIV antibody positive, active tuberculosis, HBV DNA copies>10^3/ml;
* Subjects have known or suspected brain metastases;
* Patients must receive other chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiotherapy (except for palliative local radiation) or traditional Chinese medicine for treatment of cancer during the study;
* Previously received other VEGF/VEGFR small-molecule inhibitors or antibodies therapy, including but not limited to Bevacizumab, Ramucirumab, Aflibercept;
* Previously received other HGF/c-Met small-molecule inhibitors or antibodies therapy, including but not limited to Crizotinib, Cabozantinib, Volitinib, Capmatinib (INC280), BPI-9016M;
* Imaging showed involvement of major blood vessels or nerves by tumor;
* Uncontrolled hypertension (systolic blood pressure>150mmHg and/or diastolic blood pressure>100mmHg after treatment);
* LVEF<50%;
* Apparent heart disease, including congestive heart failure(NYHA III-IV), history of myocardial infarction, or uncontrolled angina within 6 months prior to enrollment;
* Arrhythmias need to be treated, including atrial fibrillation, supraventricular tachycardia, ventricular tachycardia or ventricular fibrillation; ECG abnormalities confirmed, including QT interval prolongation (males>450msec, females>470 msec);
* History of hemorrhagic or thrombotic events within 6 months before enrollment, i.e. cerebrovascular accidents(including TIA), pulmonary embolism, spontaneous hemorrhage of tumor;
* Patients need surgery within 28 days, or is expected to require surgery within 28 days after the last dose;
* Uncontrolled cavity effusion, such as large amount of pleural effusion and ascites;
* Gastrointestinal illnesses(i.e., uncontrolled diarrhea or malabsorption) at screening or within 3 months that may affect drug absorption;
* History or suspicious signs of gastrointestinal perforation;
* Concomitant medications that may affect the drug metabolism (i.e. strong CYP3A4 inhibitors or inducer );
* Pregnant or lactating women;
* Subjects of childbearing refused to use medically acceptable methods of contraception until 3 months after the last dose;
* Participate in other clinical trials within 4 weeks prior to enrollment;
* The investigators consider the patients are not suitable for this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | until 30 days after the last dose

SECONDARY OUTCOMES:
Objective response rate | every 6 weeks, up to 2 years
Disease control rate | every 6 weeks, up to 2 years
Progression free survival | every 6 weeks, up to 2 years
Overall survival | every 6 weeks, up to 2 years
Cmax for Metatinib | day 1,day 2,day 8,day15,day22
Cmin for Metatinib | day 1,day 2,day 8,day15,day22
Tmax for Metatinib | day 1,day 2,day 8,day15,day22
AUC for Metatinib | day 1,day 2,day 8,day15,day22
T1/2 for Metatinib | day 1,day 2,day 8,day15,day22
CL for Metatinib | day 1,day 2,day 8,day15,day22

CONTACTS AND LOCATIONS:
Overall Officials: Feng Bi, MD, Principal Investigator — West China Hospital
Locations (3):
- China (3):
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang